CLINICAL TRIAL: NCT06710574
Title: Multimodal Image Technologies Investigate the Role and Mechanism of Probiotics in Improving Rapid Eye Movement Behavior Disorder with Parkinson's Disease
Brief Title: Multimodal Image Technologies Investigate the Role and Mechanism of Probiotics in Improving RBD with Parkinson's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-P2-172
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease; Movement Disorders; Rapid Eye Movement Sleep Behavior Disorder; Gut Microbiomes; Magnetic Resonance Imaging (MRI); Probiotic
Keywords: Probiotic; Parkinson's disease; Rapid Eye Movement Sleep Behavior Disorder; Multimodel Magnetic Resonance Imaging
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; REM Sleep Behavior Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- idiopathic Rapid Eye Movement sleep behavior disorder (iRBD) (Experimental): Bifidobacterium triple viable capsule (Bifico Capsule, Shanghai Shangyao Xinyi Pharmaceutical Factory Co., LTD.) 420mg, two times a day, 4 capsules each time; At the same time give the bacillus licheniformis living bacterium capsule (whole bowel capsule, northeast pharmaceutical) 0.5 g, three times a day, two at a time
  Interventions: Drug: iRBD
- Parkinson's disease without Rapid Eye Movement sleep behavior disorder (No Intervention): PD subjects without RBD matched for age and sex to PD with RBD, iRBD and healthy control subjects
- Healthy control (No Intervention): Healthy subjects without RBD matched for age and sex to PD and iRBD subjects
- Parkinson's disease with Rapid Eye Movement sleep behavior disorder group (Experimental): Bifidobacterium triple viable capsule (Bifico Capsule, Shanghai Shangyao Xinyi Pharmaceutical Factory Co., LTD.) 420mg, two times a day, 4 capsules each time; At the same time give the bacillus licheniformis living bacterium capsule (whole bowel capsule, northeast pharmaceutical) 0.5 g, three times a day, two at a time, keep the original anti Parkinson's drugs
  Interventions: Drug: PD-RBD

INTERVENTIONS:
Drug: PD-RBD — Bifidobacterium triple viable capsule (Bifico Capsule, Shanghai Shangyao Xinyi Pharmaceutical Factory Co., LTD.) 420mg, two times a day, 4 capsules each time; At the same time give the bacillus licheniformis living bacterium capsule (whole bowel capsule, northeast pharmaceutical) 0.5 g, three times a day, two at a time, keep the original anti Parkinson's drugs
  Arms: Parkinson's disease with Rapid Eye Movement sleep behavior disorder group
Drug: iRBD — Bifidobacterium triple viable capsule (Bifico Capsule, Shanghai Shangyao Xinyi Pharmaceutical Factory Co., LTD.) 420mg, two times a day, 4 capsules each time; At the same time give the bacillus licheniformis living bacterium capsule (whole bowel capsule, northeast pharmaceutical) 0.5 g, three times a day, two at a time.
  Arms: idiopathic Rapid Eye Movement sleep behavior disorder (iRBD)

SUMMARY:
Rapid eye movement sleep behavior disorder (RBD) is important non-movement feature, and also the important risk factor of Parkinson's disease (PD). In our previous work, we found that the movement features and RBD of PD patients improved after taking probiotics. The later was not reported before and the mechanism not clear. To investigate its role and mechanism, we plan to enroll patients of PD-RBD, idiopathic RBD, and healthy control, collect data of multimodal image technology before and after probiotic treatment，including resting state functional MRI，1H-MRS，123I-MIBG; analyze these data with clinical features, including UPDRS -III score, RBD-HK score , as well as the bacteria abundance and level of glutamate，GABA in blood and stool. Then, construct PD mouse model by fecal transplantation of PD patient, give or not give mouse probiotics treatment, and detect the level of glutamate, GABA, and so on, as well as α-synuclein of each brain area of each group, to explore the role and mechanism of probiotics in improving RBD and movement disorder of PD.

DETAILED DESCRIPTION:
The primary objectives of this study are to explore the effects and mechanisms of probiotic intervention on improving REM sleep behavior disorder (RBD) in patients with Parkinson's disease (PD) from both clinical and animal experimental levels. The study aims to elucidate the scientific hypothesis that "probiotic intervention improves RBD in PD patients through a neuroendocrine mechanism," providing a theoretical basis for the mechanism by which probiotic intervention alleviates RBD symptoms in PD patients.

Research Content:

Establishing imaging detection technical processes and parameters for RBD.Collecting pre- and post-probiotic treatment imaging parameters and comparing them with RBD improvement to explore the mechanism by which probiotics improve PD patient RBD.Detecting fecal microbiota abundance and blood and fecal metabolite concentrations to discuss the biochemical mechanism by which probiotics improve PD motor symptoms and RBD.

Research Methods:

Patient Recruitment:

Enrolling PD-RBD, iRBD, and healthy control subjects, with specific inclusion and exclusion criteria based on clinical diagnosis and symptomatology.

Clinical Assessments and Tests:

Utilizing standardized scales such as RBDSQ, RBD-HK, UPDRS-III, and Hoehn-Yahr staging for symptom evaluation. Conducting polysomnography (PSG) for RBD diagnosis and exclusion of other sleep disorders.

Multimodal Imaging Data Collection:

Employing 3.0T MRI for high-precision anatomical imaging, resting-state functional MRI (rs-fMRI), and proton magnetic resonance spectroscopy (1H-MRS) for glutamate, GABA, and other metabolites in specific brain regions.

Performing 123I-MIBG cardiac scintigraphy to assess cardiac sympathetic nerve function.

Laboratory Tests:

Measuring concentrations of glutamate, GABA, acetylcholine, and other metabolites in blood and fecal samples. Assessing fecal microbiota abundance through 16S rRNA gene sequencing.

Research Methods:

Patient Recruitment:

Enrolling PD-RBD, iRBD, and healthy control subjects, with specific inclusion and exclusion criteria based on clinical diagnosis and symptomatology.

Clinical Assessments and Tests:

Utilizing standardized scales such as RBDSQ, RBD-HK, UPDRS-III, and Hoehn-Yahr staging for symptom evaluation.

Conducting polysomnography (PSG) for RBD diagnosis and exclusion of other sleep disorders.

Multimodal Imaging Data Collection:

Employing 3.0T MRI for high-precision anatomical imaging, resting-state functional MRI (rs-fMRI), and proton magnetic resonance spectroscopy (1H-MRS) for glutamate, GABA, and other metabolites in specific brain regions.

Performing 123I-MIBG cardiac scintigraphy to assess cardiac sympathetic nerve function.

Laboratory Tests:

Measuring concentrations of glutamate, GABA, acetylcholine, and other metabolites in blood and fecal samples.

Assessing fecal microbiota abundance through 16S rRNA gene sequencing.

Data Analysis:

Correlating imaging data, clinical symptoms, microbiota abundance, and metabolite concentrations to explore the mechanisms of probiotic intervention in PD and RBD.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for PD-RBD patients:

* Age between 40 and 80 years, both males and females
* Patients with idiopathic Parkinson's disease, meeting the MDS clinical diagnostic criteria for Parkinson's disease (2015)
* Modified Hoehn and Yahr stage of Parkinson's disease ≤ stage 3
* No dementia, with a Mini-Mental State Examination (MMSE) score > 24
* No depression or anxiety, as indicated by Hamilton Depression Scale score < 9 and Anxiety Scale score < 14
* Rapid Eye Movement Sleep Behavior Disorder (RBD) screening questionnaire score > 5, diagnosed with RBD based on polysomnography results, and exclusion of obstructive sleep apnea
* Stable condition of Parkinson's disease motor symptoms and RBD symptoms in the month prior to enrollment, with no adjustments to Parkinson's disease medications in the month prior to enrollment
* Discontinuation of benzodiazepines such as clonazepam and melatonin in the month prior to enrollment
* No use of probiotics, prebiotics (including lactulose), or antibiotics for the two months prior to enrollment, if used, a two-month washout period should be observed
* Understanding and willingness to comply with the study protocol, agreeing to participate, and signing the informed consent form.

Inclusion criteria for iRBD patients:

* Age between 40 and 80 years, both males and females
* Rapid Eye Movement Sleep Behavior Disorder (RBD) screening questionnaire score > 5, diagnosed with RBD based on polysomnography results, and exclusion of obstructive sleep apnea or restless legs syndrome
* No dementia, with a Mini-Mental State Examination (MMSE) score > 24
* No depression or anxiety, as indicated by Hamilton Depression Scale score < 9 and Anxiety Scale score < 14
* Discontinuation of benzodiazepines such as clonazepam and melatonin in the month prior to enrollment
* No use of probiotics, prebiotics (including lactulose), or antibiotics for the two months prior to enrollment, if used, a two-month washout period should be observed
* Understanding and willingness to comply with the study protocol, agreeing to participate, and signing the informed consent form.

Inclusion criteria for healthy subjects

* Age between 40 and 80 years, age and gender matched with the above two groups of patients
* Rapid Eye Movement Sleep Behavior Disorder screening questionnaire score ≤ 5, exclusion of RBD or obstructive sleep apnea based on polysomnography results
* No dementia, with a Mini-Mental State Examination (MMSE) score > 24.
* No depression or anxiety, as indicated by Hamilton Depression Scale score < 9 and Anxiety Scale score < 14
* No severe constipation, not meeting the diagnostic criteria for Rome III chronic constipation; No use of probiotics, prebiotics (including lactulose), or antibiotics for the two months prior to enrollment, if used, a two-month washout period should be observed
* Understanding and willingness to comply with the study protocol, agreeing to participate, and signing the informed consent form.

Exclusion Criteria:

PD-RBD exclusion criteria:

* Parkinsonism plus syndrome and secondary parkinsonism such as multiple system atrophy, progressive supranuclear palsy, cortical basal ganglia degeneration, dementia with Lewy bodies, vascular parkinsonism, post-encephalitis parkinsonism, or any other non-primary parkinsonism
* Taking any probiotics or prebiotics (including lactulose) or antibiotics within 2 months before enrollment
* Adjustment of Parkinson's disease medication within 1 month before enrollment; In group 1 month before taking clonazepam and benzodiazepines medicine melatonin, etc.
* With the following diseases such as Alzheimer's disease, malignant tumor, spinal cord lesions, epilepsy, autonomic nerve disease (urinary retention, urinary incontinence or orthostatic hypotension, vertical drop in blood pressure in five minutes more than 30/15 MMHG), etc.; New onset of cerebrovascular disease or severe sequelae of cerebrovascular disease within 3 months, affecting the assessment
* Patients with anxiety or depression and taking medication
* Serious cardiovascular diseases (such as the American heart association heart function class for Ⅲ - Ⅳ of congestive heart failure, the 6 month history of myocardial infarction, etc.)
* Severe liver and kidney dysfunction, cereal third transaminase, aspertate aminotransferase, total bilirubin is higher than the upper limit of normal value of 1. 5 times; Serum creatinine is higher than the upper limit of normal value 1. 5 times
* Pregnant and lactating women or pregnant women aged 40-60 years with positive HCG;
* Known to be allergic to Bifidobacterium triple viable capsules, Bacillus licheniformis, or their excipients
* Has a history of history of drug abuse or alcohol dependence
* Were enrolled in another clinical trial at enrollment
* Refusal to participate in the study or inability to cooperate with the study investigator; The researchers judgment for doesn't fit into the group of patients.

Exclusion criteria for iRBD:

* PD motor symptoms and parkinsonism were included in the PD-RBD group; "Parkinsonism plus syndrome and secondary parkinsonism, such as multiple system atrophy, progressive supranuclear palsy, cortical basal ganglia degeneration, dementia with Lewy bodies, vascular parkinsonism, post-encephalitis parkinsonism, or any other non-primary Parkinson's disease;"
* Into the group 2 months before taking any probiotics and prebiotics (including lactulose) or antibiotics
* Adjustment of Parkinson's disease medication within 1 month before enrollment; In group 1 month before taking clonazepam and benzodiazepines medicine melatonin, etc.
* With the following diseases, including but not limited to obstructive sleep apnea syndrome, Alzheimer disease, malignant tumor, spinal cord lesions, epilepsy, autonomic nerve disease (urinary retention, urinary incontinence or orthostatic hypotension, vertical drop in blood pressure in five minutes more than 30/15 MMHG), etc.; 3 month new cerebrovascular disease or severe cerebrovascular disease sequela, impact assessment;
* Patients with severe anxiety or depression or under drug treatment;
* Severe cardiovascular diseases (such as congestive heart failure with American Heart Association functional class Ⅲ-Ⅳ, history of myocardial infarction within 6 months, etc.);
* Severe liver and kidney dysfunction, cereal third transaminase, aspertate aminotransferase, total bilirubin is higher than the upper limit of normal value of 1. 5 times; The serum creatinine was higher than the upper limit of the normal range. 5 times;
* Pregnant and lactating women or pregnant women aged 40-60 years with positive HCG;
* Known to be allergic to Bifidobacterium triple viable capsules, Bacillus licheniformis, or their excipients;
* With a history of drug abuse or alcohol dependence
* Were enrolled in another clinical trial at enrollment;
* Refused into groups, and can cooperate with researchers; Patients who were judged by the investigator to be ineligible for enrollment.

Healthy subjects exclusion criteria:

* Patients with Parkinson's disease motor symptoms and met the diagnosis of parkinsonism were included in PD-RBD group; "Parkinsonism plus syndrome and secondary parkinsonism, such as multiple system atrophy, progressive supranuclear palsy, cortical basal ganglia degeneration, dementia with Lewy bodies, vascular parkinsonism, post-encephalitis parkinsonism, or any other non-primary Parkinson's disease;" 2) taking any probiotics or prebiotics (including lactulose) or antibiotics within 2 months before enrollment; 1 month before the 3) into the group of Parkinson's disease medication adjustment; Benzodiazepines such as clonazepam and melatonin were taken within 1 month before enrollment. 4) combined with the following diseases, including but not limited to obstructive sleep apnea syndrome, Alzheimer's disease, malignant tumors, spinal cord lesions, epilepsy, autonomic disorders (urinary retention, urinary incontinence or orthostatic hypotension, blood pressure drop more than 30/15 MMHG after 5 minutes of standing), etc.; New onset of cerebrovascular disease or severe sequelae of cerebrovascular disease within 3 months, affecting the assessment
* Patients with severe anxiety or depression or under drug treatment;
* Severe cardiovascular diseases (such as congestive heart failure with American Heart Association functional class Ⅲ-Ⅳ, history of myocardial infarction within 6 months, etc.)
* Severe liver and kidney dysfunction, cereal third transaminase, aspertate aminotransferase, total bilirubin is higher than the upper limit of normal value of 1. 5 times; The serum creatinine was higher than the upper limit of the normal range. 5 times
* Pregnant and lactating women or pregnant women aged 40-60 years with positive HCG; 9) known to the bifidobacterium triple viable capsules, bacillus licheniformis, or its accessories, and other allergies;
* With a history of drug abuse or alcohol dependence
* Were enrolled in another clinical trial at enrollment;
* Refused into groups, and can cooperate with researchers; The researchers judgment for doesn't fit into the group of patients.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Magnetic resonance imaging changes of brain structure and function | 12 weeks
Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale(MDS-UPDRS) | 12 weeks
The abundance of gut microbiota | 12 weeks

SECONDARY OUTCOMES:
Patient assessment of constipation symptom | 12 weeks
Epworth sleepiness score | 12 weeks
Hoehn-Yahr | 12 weeks
RBD Questionnaire-Hong Kong | 12 weeks
Rapid-eye-movement Sleep Behavior Disorder Screening Questionnaire | 12 weeks
Pittsburgh Sleep Quality Index | 12 weeks
Cleveland Clinic Score | 12 weeks
Functional constipation diagnostic standard scale | 12 weeks
Glutamate (blood) | 12 weeks
Glutamate (feces) | 12 weeks
N-acetylaspartate(blood) | 12 weeks
N-acetylaspartate(feces) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valencia Garcia S, Libourel PA, Lazarus M, Grassi D, Luppi PH, Fort P. Genetic inactivation of glutamate neurons in the rat sublaterodorsal tegmental nucleus recapitulates REM sleep behaviour disorder. Brain. 2017 Feb;140(2):414-428. doi: 10.1093/brain/aww310. Epub 2016 Dec 21. PMID 28007991
- [Background] Henrich MT, Geibl FF, Lee B, Chiu WH, Koprich JB, Brotchie JM, Timmermann L, Decher N, Matschke LA, Oertel WH. A53T-alpha-synuclein overexpression in murine locus coeruleus induces Parkinson's disease-like pathology in neurons and glia. Acta Neuropathol Commun. 2018 May 10;6(1):39. doi: 10.1186/s40478-018-0541-1. PMID 29747690
- [Background] Knudsen K, Fedorova TD, Hansen AK, Sommerauer M, Otto M, Svendsen KB, Nahimi A, Stokholm MG, Pavese N, Beier CP, Brooks DJ, Borghammer P. In-vivo staging of pathology in REM sleep behaviour disorder: a multimodality imaging case-control study. Lancet Neurol. 2018 Jul;17(7):618-628. doi: 10.1016/S1474-4422(18)30162-5. Epub 2018 Jun 1. PMID 29866443
- [Background] Pyatigorskaya N, Gaurav R, Arnaldi D, Leu-Semenescu S, Yahia-Cherif L, Valabregue R, Vidailhet M, Arnulf I, Lehericy S. Magnetic Resonance Imaging Biomarkers to Assess Substantia Nigra Damage in Idiopathic Rapid Eye Movement Sleep Behavior Disorder. Sleep. 2017 Nov 1;40(11). doi: 10.1093/sleep/zsx149. PMID 28958075
- [Background] Mayer G, Bitterlich M, Kuwert T, Ritt P, Stefan H. Ictal SPECT in patients with rapid eye movement sleep behaviour disorder. Brain. 2015 May;138(Pt 5):1263-70. doi: 10.1093/brain/awv042. Epub 2015 Mar 1. PMID 25732183
- [Background] Rahayel S, Postuma RB, Montplaisir J, Bedetti C, Brambati S, Carrier J, Monchi O, Bourgouin PA, Gaubert M, Gagnon JF. Abnormal Gray Matter Shape, Thickness, and Volume in the Motor Cortico-Subcortical Loop in Idiopathic Rapid Eye Movement Sleep Behavior Disorder: Association with Clinical and Motor Features. Cereb Cortex. 2018 Feb 1;28(2):658-671. doi: 10.1093/cercor/bhx137. PMID 28591814
- [Background] De Marzi R, Seppi K, Hogl B, Muller C, Scherfler C, Stefani A, Iranzo A, Tolosa E, Santamaria J, Gizewski E, Schocke M, Skalla E, Kremser C, Poewe W. Loss of dorsolateral nigral hyperintensity on 3.0 tesla susceptibility-weighted imaging in idiopathic rapid eye movement sleep behavior disorder. Ann Neurol. 2016 Jun;79(6):1026-30. doi: 10.1002/ana.24646. Epub 2016 Apr 22. PMID 27016314
- [Background] Rolinski M, Griffanti L, Piccini P, Roussakis AA, Szewczyk-Krolikowski K, Menke RA, Quinnell T, Zaiwalla Z, Klein JC, Mackay CE, Hu MT. Basal ganglia dysfunction in idiopathic REM sleep behaviour disorder parallels that in early Parkinson's disease. Brain. 2016 Aug;139(Pt 8):2224-34. doi: 10.1093/brain/aww124. Epub 2016 Jun 12. PMID 27297241
- [Background] Luppi PH. Jouvet's animal model of RBD, clinical RBD, and their relationships to REM sleep mechanisms. Sleep Med. 2018 Sep;49:28-30. doi: 10.1016/j.sleep.2018.05.026. Epub 2018 Jun 6. PMID 30172630
- [Background] Alam R, Abdolmaleky HM, Zhou JR. Microbiome, inflammation, epigenetic alterations, and mental diseases. Am J Med Genet B Neuropsychiatr Genet. 2017 Sep;174(6):651-660. doi: 10.1002/ajmg.b.32567. Epub 2017 Jul 10. PMID 28691768
- [Background] Fang X. Potential role of gut microbiota and tissue barriers in Parkinson's disease and amyotrophic lateral sclerosis. Int J Neurosci. 2016 Sep;126(9):771-6. doi: 10.3109/00207454.2015.1096271. Epub 2015 Oct 16. PMID 26381230
- [Background] Stolzenberg E, Berry D, Yang D, Lee EY, Kroemer A, Kaufman S, Wong GCL, Oppenheim JJ, Sen S, Fishbein T, Bax A, Harris B, Barbut D, Zasloff MA. A Role for Neuronal Alpha-Synuclein in Gastrointestinal Immunity. J Innate Immun. 2017;9(5):456-463. doi: 10.1159/000477990. Epub 2017 Jun 27. PMID 28651250
- [Background] Sampson TR, Debelius JW, Thron T, Janssen S, Shastri GG, Ilhan ZE, Challis C, Schretter CE, Rocha S, Gradinaru V, Chesselet MF, Keshavarzian A, Shannon KM, Krajmalnik-Brown R, Wittung-Stafshede P, Knight R, Mazmanian SK. Gut Microbiota Regulate Motor Deficits and Neuroinflammation in a Model of Parkinson's Disease. Cell. 2016 Dec 1;167(6):1469-1480.e12. doi: 10.1016/j.cell.2016.11.018. PMID 27912057
- [Background] Scheperjans F, Aho V, Pereira PA, Koskinen K, Paulin L, Pekkonen E, Haapaniemi E, Kaakkola S, Eerola-Rautio J, Pohja M, Kinnunen E, Murros K, Auvinen P. Gut microbiota are related to Parkinson's disease and clinical phenotype. Mov Disord. 2015 Mar;30(3):350-8. doi: 10.1002/mds.26069. Epub 2014 Dec 5. PMID 25476529